CLINICAL TRIAL: NCT05143346
Title: A Comparison Between Using Video Stylet and Video Laryngoscope in Difficult Intubation of Traumatic Patients .
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, WTMahran, Doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Difficult intubation
Record Dates: First submitted 2021-10-23; First posted 2021-12-03 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Difficult or Failed Intubation
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Other): Group A will include 33 patients and will be intubated by the use of video stylet.
  Interventions: Device: Intubation
- Group B (Other): Group B will include 33 patients and will intubated by the use of video laryngoscope
  Interventions: Device: Intubation

INTERVENTIONS:
Device: Intubation — Using video stylet and video laryngoscope in difficult intubation in patients with trauma or suspected to be have difficult intubation.

SUMMARY:
The aim of this study is to compare the visualization of the glottis, the time for tracheal intubation, the success rate of intubation, and the need for manoeuvres to optimize the view using video stylet or video laryngoscope in patients with expected difficult intubations.

DETAILED DESCRIPTION:
The airway, breathing and circulation support '' ABCs" of trauma resuscitation were born from the assumption that correcting hypoxemia and hypotension reduces morbidity and mortality. Definitive care for severely injured or polytrauma patients includes the ability to provide advanced airway management in a variety of settings: in the emergency department, 20% to 30% intubations are for trauma. Airway management in traumatic patient presents numerous unique challenges beyond placement of an endotracheal tube, without comes dependent on the provider's ability to predict and anticipate difficulty and have a safe and executable plan. In severely injured patients, the cervical spine must be protected by in-line immobilisation during airway management. If orotracheal intubation is required, then manual in-line stabilisation is recommended to facilitate tracheal intubation to secure a space for tongue displacement into the submandibular space. However, manual in-line stabilisation can make alignment of the oral, pharyngeal and laryngeal axes difficult, resulting in a poor direct laryngoscopic view and prolonging the intubation time. Video stylets, which are portable and easier to prepare than flexible fiberoptic bronchoscopes, could be better option for tracheal intubation in patient with cervical immobilization. Previous studies have shown the usefulness of video stylets for tracheal intubation in cervical immobilized patients.

Video laryngoscopes provide a better laryngeal view. They are easy to use and have a high success rate and short intubation time in patients with predicted difficult airways. Successful use of video laryngoscopy is increasing for airway management of patients with trauma in the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Any patient in the age group of (5 - 80) and has
* Suspected difficult intubation.
* High mallampati score (class 111, 1V).
* Suspected cervical fracture.
* Maxillofacial trauma.
* Fracture base of the skull.
* Polytrauma.

Exclusion Criteria:

* Patients with low mallampati score (class 1, 11).
* Patients undergoing elective surgeries and not suspected to have difficult intubations.
* Patients aged below 5 years and above 80 years.

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Comparison of success rate for the tracheal intubation in patients with anticipated difficult airways, demonstrating the non inferiority of video stylet efficacy compare to the most consolidated technique based on videolaryngoscope | 5 minutes
  The success rate of the rigid fiberoptic stylet to perform tracheal intubation in patients with anticipated difficult airways [ Time Frame: up to a maximum of 3 attempts and up to 3 minutes from device insertion for each attempt (max 3 minutes) ]
  .
  success rate of the procedure defined as correct positioning of the tracheal tube in the trachea confirmed both endoscopically and through the capnographic curve end tidal carbon dioxide (Et CO2) time consumed to achieve a successful intubation by each device.

SECONDARY OUTCOMES:
Average time of intubation procedure expressed in seconds [ Time Frame: up to 3 minutes ] | 3 minutes
  Time in minutes measured from device insertion into the patient's mouth until the endotracheal tube will be positioned into the trachea
  .
Development of any complications [ Time Frame: up to 6 hours measured from the insertion of the device ] | 6 hours
  Occurrence of any complications or adverse event during the procedure (desaturation episodes, hemodynamic changes, oral-pharynx and larynx traumatism)

CONTACTS AND LOCATIONS:
Locations (1):
- Wesam Mahran, Asyut, Egypt

REFERENCES:
- [Background] Tosone SR, Reves JG, Kissin I, Smith LR, Fournier SE. Hemodynamic responses to nifedipine in dogs anesthetized with halothane. Anesth Analg. 1983 Oct;62(10):903-8. PMID 6614523
- [Background] Hayat K, Finnegan M, Lee KA, Rees RC, Hancock BW, Goyns MH. Variable expression of the interleukin-2 receptor alpha chain and MYC genes in lymphocytes from renal cell carcinoma patients treated with interleukin-2. Cancer Lett. 1992 Aug 14;65(2):173-8. doi: 10.1016/0304-3835(92)90163-p. PMID 1511423